CLINICAL TRIAL: NCT03706911
Title: An Open-label Study to Evaluate Safety, Tolerability and Pharmacokinetics of VM-1500A-LAI After Single and Multiple Ascending Dose Administration to Healthy Volunteers
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of VM-1500A-LAI Single and Multiple Ascending Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HIV-VM1500ALAI-01
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: HIV-1-infection
Keywords: HIV-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- VM-1500A-LAI 150mg (Experimental): VM-1500A-LAI 150mg IM single dose
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI 300mg (Experimental): VM-1500A-LAI 300mg IM single dose
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI 600mg (Experimental): VM-1500A-LAI 600mg IM single dose
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI 1200mg (Experimental): VM-1500A-LAI 1200mg IM single dose
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI 600 mg Multiple (Experimental): VM-1500A-LAI Multiple dose (2 injections every 4 weeks)
  Interventions: Drug: VM-1500A-LAI

INTERVENTIONS:
Drug: VM-1500A-LAI — VM-1500A (parent drug of elsulfavirine) IM injection dosage form
  Other Names: VM-1500; VM-1500A

SUMMARY:
To evaluate safety and tolerability of VM-1500A-LAI after its single and multiple intramuscular ascending dose to healthy volunteers

DETAILED DESCRIPTION:
Primary Objective:

To evaluate safety and tolerability of VM-1500A-LAI after its single and multiple intramuscular ascending dose to healthy volunteers.

Secondary Objectives:

To evaluate pharmacokinetic parameters of VM-1500A after its single and multiple intramuscular ascending dose administration to healthy volunteers.

To evaluate safety and tolerability of ELPIDA®, administered in the run-in period

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking healthy male subjects aged 18 - 45 years (inclusive);
2. Verified "healthy" status, based on standard clinical, laboratory, and instrumental examination methods;
3. Body weight ≥ 50 kg and Body Mass Index in the range from 18.5 to 30.0 kg/m2;
4. Signed the Participant Explanation Sheet and the Informed Consent Form;
5. Consent to use an adequate method of contraception throughout the study and 3 months after its completion: a condom with spermicide substance (cream, foam or suppository).

Exclusion Criteria:

1. Chronic cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal or gastrointestinal diseases, as well as immunologic, hepatic, renal, or blood diseases;
2. Laboratory abnormalities, or ECG abnormalities at Screening;
3. Systolic arterial pressure less than 90 mm Hg or above 130 mm Hg, diastolic arterial pressure less than 60 mm Hg or above 85 mm Hg, heart rate less than 60 BPM or more than 90 BPM at Screening;
4. Regular intake of drugs within 2 weeks before Screening (including herbal preparations and dietary supplements); intake of drugs that have a pronounced effect on hemodynamics, liver, kidney, or CNS function, etc. (for example, barbiturates, omeprazole, cimetidine, etc.) within 4 weeks before Screening;
5. Presence of antibodies to HIV or hepatitis C virus, presence of hepatitis В surface antigen, positive syphilis test;
6. Unstable sleeping (for example, night work, sleep disturbances, insomnia, recent return from another time zone, etc.);
7. Signs of alcohol (taking more than 10 units of alcohol per week) or drug addiction; alcohol or drugs consumption within 7 days prior to Screening; smoking within 3 months before Screening; positive drug or alcohol test at Screening;
8. Depression episodes or other mental disorders/conditions in medical history that required therapy
9. Allergy in medical history (including drug intolerance and food allergy);
10. Hypersensitivity to the active substance or to any other ingredient of the study drug. Sucrose intolerance, sucrase-isomaltase deficiency, sucrose isomaltose malabsorption, lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
11. Blood/plasma donation (450 ml or more of blood/plasma) or surgical intervention within 12 months before Screening;
12. Diseases and conditions (current or in medical history), including surgical intervention, which, according to the opinion of Investigator, may affect the absorption, distribution, metabolism, or excretion of the study drug (excluding appendectomy);
13. Participation in other clinical studies or therapy with other study drugs within 3 months before Screening;
14. Acute infectious diseases within 4 weeks before Screening;
15. Subjects unable to read or write; unwillingness to understand and follow to the procedures, defined in the Study Protocol; non-compliance with the dosing regimen or procedures, which according to the opinion of Investigator, may affect the study results or safety of study subject and prevent the subject from further participation in the study; any other associated medical or serious mental conditions making the subject not eligible to participate in the clinical study, restricting validity of obtaining the informed consent or affecting the subject's ability to participate in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male volunteers will be included in this study
Enrollment: 27 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
The incidence of AEs and SAEs. Concentration of VM1500A in plasma and RBCs | 4 weeks for SAD, 8 weeks for MAD
  The incidence of adverse events (AEs) and serious adverse events (SAEs). This is an open-label study aimed to evaluate safety, tolerability, and pharmacokinetics of VM-1500A-LAI administered as single or multiple ascending doses to healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Smolyarchuk, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No